CLINICAL TRIAL: NCT05347992
Title: ELEVATE - (Empower Lupus Erythematosus Patients Via Allowing RemoTe Evaluation)
Acronym: ELEVATE
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: DXT-MCD-AI01
Record Dates: First submitted 2022-04-11; First posted 2022-04-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fingerstick blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care: Cohort(1) of the study will collect longitudinal blood samples from participants who are on the standard of care treatment for Systemic lupus erythematosus (SLE) based on Cohort specific inclusion criteria
- Biologics: Cohort(2) of the study will collect longitudinal blood samples from participants who are on biologics treatment for Systemic lupus erythematosus (SLE) based on Cohort specific inclusion criteria

SUMMARY:
To explore the potential for use of DxTerity's AIP IFN-1 test as personalized guided care and monitoring module in patients with Systemic lupus erythematosus(SLE) using consented patient health information

DETAILED DESCRIPTION:
Explore and demonstrate concordance between self-collected samples and traditional phlebotomist venous draw for DxTerity AIP module and biomarkers like C3, C4, anti dsDNA and CRP in SLE participants with self-reported outcomes and medical record data.

The study will collect blood samples and self-reported information for SLE subjects, up to 5000 participants in Phase I, with a subset of 1000 continuing to Phase II with Medical records. Study participants will be recruited using a combination of digital media (including social media, advertising, bloggers, emails). Enrollment and qualification will be done along with consented retrieval of medical records using a study specific mobile app.

ELIGIBILITY:
Inclusion Criteria: (PHASE I)

1. Individuals aged 18 years or older.
2. Must reside in United States
3. Have a clinical diagnosis of SLE
4. Willingness to consent to provide electronic medical records (EMR)
5. Provide written informed consent and comply with the study procedures.

(PHASE II)

1. Verified diagnosis (Medical records or /and Physician Questionnaire) for SLE
2. Report one or more of the following (record all that apply):

   1. Worsening or changes in symptoms or flare
   2. Changes in treatment regimen
   3. On standard of care treatment
   4. On biologics

Exclusion Criteria:

1. Participants unable to complete study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with SLE
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Concordance between self collected samples and traditional venous draws | 36 months
  Percentage of participants with concordant IFN-1 status as assessed by the DxTerity AIP IFN-1 module, concordance between phlebotomy draw and self-collected blood samples.

SECONDARY OUTCOMES:
Longitudinal monitoring | 36 months
  Percentage of participants with correlation between IFN-1 high status and increased flares by SAF36 and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Terbrueggen, PhD, Principal Investigator — DxTerity Diagnostics
Locations (1):
- DxTerity Diagnostics, Inc., Compton, California, United States

IPD SHARING:
Plan to Share IPD: No